CLINICAL TRIAL: NCT01222975
Title: Single Dose Two-way Crossover Fasted Bioequivalence Study of Risperidone 1 mg ODT Tablets in Healthy Volunteers
Brief Title: Bioequivalence Study of Risperidone 1 mg Orally-disintegrating Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AAI-US-257
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: risperidone fasting study
MeSH Terms: interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Risperidone orally disintegrating tablets of Ranbaxy Laboratories, Ltd
  Interventions: Drug: Risperidone
- 2 (Active Comparator): Risperdal® M-Tab of Janssen Pharmaceutica Products L.P.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — orally disintegrating tablets

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and bioequivalence of Risperidone formulations after administration of single doses to normal, healthy subjects under fasted conditions.

DETAILED DESCRIPTION:
A single dose two way crossover bioequivalence study in 44 normal healthy males and females was utilized to evaluate the pharmacokinetics and bioequivalence of Risperidone ODT (orally dissolving tablet) formulations. The test product was a 1 mg ODT tablet formulation of Risperidone manufactured by Ranbaxy Laboratories Ltd. The reference product was commercially available Risperidone 1 mg ODT tablets (Risperdal®), Janssen Pharmaceutica Products, LP. Each single oral dose (1 mg) will be administered orally as a 1 mg tablet. Blood samples were collected at intervals over a 72-hour period after medication administration. There was a washout period of 14 days between the two periods of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects at least 18 years of age
2. Informed of the nature of the study and given written informed consent
3. Have a body weight within 15% of the appropriate range as defined in the 1983 Metropolitan Life Company tables weighing at least 110 pounds

Exclusion Criteria:

1. Hypersensitivity to risperidone (Risperdal®)
2. Any history of a clinical condition that might affect drug absorption, metabolism or excretion
3. Recent history (within one year) of mental illness, drug addiction, drug abuse or alcoholism
4. Donation of greater than 500 mg of blood in the past 4 weeks prior to study dosing or difficulty in donating blood
5. Received an investigational drug within the 4 weeks prior to study dosing
6. Currently taking any prescription medication, except for oral contraceptives, within the 7 days prior to the study dosing or over the counter medication within 3 days of study dosing. This prohibition does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physician
7. Regular smoking or more than 5 cigarettes daily or the daily use of nicotine-containing products beginning 3 months before the study medication administration through the final evaluation
8. If female the subject is lactating or has a positive pregnancy test at screening and prior to each of the treatment periods. Females of child-bearing potential must use a medically acceptable method of contraception throughout the study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/ or her partner are: oral contraceptives, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization of their partner(s) or abstinence. Females taking oral contraceptives must have taken them consistently for at least three months prior to receiving study medication
9. Alcohol, grapefruit beverages or foods or caffeine beverages or foods beginning 1 days before each study medication administration through each study confinement period. Such restricted items include coffee, tea, iced tea, coke®, Pepsi®, mountain dew®, chocolate, brownies, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-10; Primary Completion 2004-10 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of Risperidone 1 mg Orally-disintegrating tablets

CONTACTS AND LOCATIONS:
Locations (1):
- aaiPharma Inc., Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html
- See also: Related Info — http://www.fda.gov/Safety/Recalls/default.htm
- See also: Related Info — http://www.fda.gov/Safety/MedWatch/default.htm